CLINICAL TRIAL: NCT02636049
Title: Pharmacokinetics of Triferic (Ferric Pyrophosphate Citrate) Administered Intravenously to Healthy Adult Volunteers
Acronym: RMFPC-12
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-12
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: End Stage Renal Disease
Keywords: pharmacokinetics; healthy adult volunteer
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Period: 6 mg Triferic IV over 3 hours (Experimental): Each subject will receive a single 6 mg dose of Triferic administered as a continuous intravenous infusion over 3 hours on Day 2. The Triferic IV dosing solution will have been prepared by diluting Triferic from ampules (5.44 mg/mL) in an appropriate amount of D5W to a concentration of 0.020 mg/mL. Administration of 300 mL IV at 100 mL/hr for 3 hours results in delivery of 6 mg of Triferic iron.
  Interventions: Drug: Triferic
- Treatment Period: 35 micrograms/kg IV push (Experimental): Each subject will receive Triferic as 35 µg/kg body weight IV push over 30-60 seconds on Day 3. The Triferic IV push dosing solution will have been prepared by diluting Triferic from ampules (5.44 mg/mL) in an appropriate amount of D5W to a concentration of 35 µg Triferic iron/kg body weight per subject in 4.5 mL.
  Interventions: Drug: Triferic

INTERVENTIONS:
Drug: Triferic — Triferic is supplied as sterile 5 mL ampules containing 5.44 mg/mL of iron in water for injection. Each 5 mL ampule contains 27.2 mg of Triferic iron.
  Other Names: ferric pyrophosphate citrate; FPC

SUMMARY:
This is a Phase 1, open-label, three-period sequential dosing study being conducted to determine the pharmacokinetics of Triferic iron administered intravenously (IV) to healthy adults.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, three-period sequential dosing study being conducted primarily to determine the pharmacokinetics of Triferic iron administered intravenously to healthy adults.. Participation will be up to 5 weeks total duration including Screening, Baseline, Treatment Period, and Follow-up. Following Screening, subjects will be admitted to the clinic on Day -1, prior to Baseline (Day 1). During the Treatment Period, subjects will receive two doses of Triferic. Each subject will receive a single 6-mg dose of Triferic administered IV over 3 hours (hr) on one day (Day 2), and a single 35-µg/kg dose of Triferic administered IV push the following day (Day 3). On Day 4, subjects will be discharged from the clinic and will return approximately one week later for their final Follow-up visit.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following criteria to be eligible for inclusion in the study:

1. The subject must be able to provide informed consent and have personally signed and dated the study written informed consent document before completing any study-related procedures.
2. The subject must be 18-65 years of age inclusive at the time of consent.
3. The subject must have a transferrin saturation (TSAT) of 15-50% during Screening.
4. The subject must agree to discontinue all iron preparations for 14 days prior to Baseline.
5. If the subject is female, she must be premenopausal, non-pregnant and non-lactating, and be at least 90 days post-partum (if applicable) at Screening. Women of childbearing potential must be willing to use appropriate birth control during the entire duration of the study.
6. The subject must be willing and able to comply with all study procedures and restrictions.
7. The subject must have no clinically-significant abnormal findings on medical history, vital signs, physical examination, or clinical laboratory results during Screening.
8. The subject must have a body mass index (BMI) of ≤32.0 kg/m2 at Screening and weigh >60.0 kg.

Exclusion Criteria:

A subject will not be eligible for inclusion in the study if any of the following criteria apply:

1. The subject has a hemoglobin (Hgb) concentration <13.0 g/dL for men or <12 g/dL for women during Screening.
2. The subject has a total iron binding capacity (TIBC) <250 µg/dL during Screening.
3. The subject has had administration of IV or oral iron supplements (including multivitamins with iron) within 14 days prior to Baseline.
4. Subject has concurrent or recurrent disease (e.g., cardiovascular, renal, hepatic, gastrointestinal, malignant, etc.) that could affect the action or disposition of the investigational product utilized in this study, or could affect clinical or laboratory assessments.
5. Subject has a C-reactive protein level (CRP) >5 mg/L during Screening, or any rheumatic or autoimmune disease that requires systemic anti-inflammatory or immunomodulatory therapy.
6. Subject has an acute illness within 14 days prior to Baseline.
7. Subject has known or suspected intolerance or hypersensitivity to iron-containing products.
8. Subject has a history of alcohol or substance abuse within the past year.
9. Subject has a positive screen for cotinine or drugs of abuse.
10. Subject is positive for HIV, hepatitis B, or hepatitis C.
11. Subject uses tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, etc.). Ex-users must report that they have stopped using tobacco for at least 30 days prior to Baseline.
12. Subject donated blood or blood products (e.g., plasma or platelets) within 60 days prior to Baseline.
13. Subject participated in an investigational drug study within 30 days prior to Baseline.
14. Subject is pregnant or intends to become pregnant before completing the study.
15. Subject's current medical status, in the investigator's opinion, would preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD FACP, Study Director — Rockwell Medical, Inc
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: After enrollment, all subjects underwent blood sampling for pharmacokinetic (PK) purposes over 16 hours on Day 1 to establish a baseline. On Day 2, subjects received a single 6 mg dose of Triferic administered as a continuous intravenous infusion over 3 hours, with blood sampling for PK purposes over 16 hours. On Day 3, subject received Triferic 35 micrograms/kg as an intravenous push (administered in 30 - 60 seconds), with blood sampling for PK purposes over 16 hours.
  Triferic: Triferic is supplied as sterile 5 mL ampules containing 5.44 mg/mL of iron in water for injection. Each 5 mL ampule contains 27.2 mg of Triferic iron.
Period: Overall Study
Arm/Group | All Participants
Started | 12
Triferic 6 mg IV Over 3 Hours | 12
Triferic 35 Micrograms/kg IV Push | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All 12 participants completed every arm of the study. Therefore, the baseline demographic characteristics of the Safety Population as a whole also reflect the characteristics of each arm of the study.
Arm/Group | Safety Population
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Height [Mean (Standard Deviation); unit: centimeters] | 179.61 (7.365)
Weight [Mean (Standard Deviation); unit: kilogram] | 84.48 (12.892)
Body Mass Index [Mean (Standard Deviation); unit: Kilogram/square meter] | 26.07 (2.592)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Triferic Iron Administered IV to Healthy Adults: Maximum Drug Concentration (Cmax) of Total Serum Iron
Description: Blood samples will be drawn at time = 0, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12, and 16 hours after the start of Triferic administration on study Day 2 (IV infusion of 6 mg Triferic over 3 hours) and Day 3 (35 microgram/kg IV dose of Triferic given over 30 - 60 seconds) in order to determine the Peak Serum Concentration, corrected (Cmax) of total serum iron.
Time Frame: 16 hours
Population: Pharmacokinetic population: all enrolled subjects who received at least 1 dose of study drug and had sufficient pharmacokinetic samples (a sample at the end of infusion and at least 3 samples during the elimination phase) for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/deciliter
Groups:
- Treatment Period: 6 mg Triferic IV Over 3 Hours: Each subject will receive a single 6 mg dose of Triferic administered as a continuous intravenous infusion over 3 hours. The Triferic IV dosing solution will have been prepared by diluting Triferic from ampules (5.44 mg/mL) in an appropriate amount of D5W to a concentration of 0.020 mg/mL. Administration of 300 mL IV at 100 mL/hr for 3 hours results in delivery of 6 mg of Triferic iron.
  Triferic: Triferic is supplied as sterile 5 mL ampules containing 5.44 mg/mL of iron in water for injection. Each 5 mL ampule contains 27.2 mg of Triferic iron.
- Treatment Period: 35 Micrograms/kg IV Push: Each subject will receive Triferic as 35 µg/kg body weight IV push over 30-60 seconds. The Triferic IV push dosing solution will have been prepared by diluting Triferic from ampules (5.44 mg/mL) in an appropriate amount of D5W to a concentration of 35 µg Triferic iron/kg body weight per subject in 4.5 mL.
  Triferic: Triferic is supplied as sterile 5 mL ampules containing 5.44 mg/mL of iron in water for injection. Each 5 mL ampule contains 27.2 mg of Triferic iron.
Arm/Group | Treatment Period: 6 mg Triferic IV Over 3 Hours | Treatment Period: 35 Micrograms/kg IV Push
Number analyzed (Participants) | 11 | 12
microgram/deciliter | 102 (40.1) | 44.1 (71.9)

2. Primary Outcome: Pharmacokinetics of Triferic Iron Administered IV to Healthy Adults: Area Under the Serum Iron Concentration Time Curve From Time Zero to the Time of Last Quantified Concentration (AUC(Last)) of Total Serum Iron
Description: Blood samples will be drawn at time = 0, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12, and 16 hours after the start of Triferic administration on study Day 2 (IV infusion of 6 mg Triferic over 3 hours) and study day 3 (35 microgram/kg IV Triferic dose administered in 30 - 60 seconds) in order to determine the AUC(last) of total serum iron.
Time Frame: 16 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/deciliter
Arm/Group | Treatment Period: 6 mg Triferic IV Over 3 Hours | Treatment Period: 35 Micrograms/kg IV Push
Number analyzed (Participants) | 11 | 12
hour*microgram/deciliter | 858 (59.6) | 175 (234)

3. Secondary Outcome: Incidence of Treatment Emergent Adverse Events
Description: The number of patients that experienced treatment emergent adverse events will be quantified.
Time Frame: 10 - 14 days
Population: Safety Population: all enrolled subjects
Measure: Number; unit: participants
Arm/Group | Treatment Period: 6 mg Triferic IV Over 3 Hours | Treatment Period: 35 Micrograms/kg IV Push
Number analyzed (Participants) | 12 | 12
participants | 1 | 1

4. Secondary Outcome: Incidence of Treatment Emergent Serious Adverse Events
Description: The number of patients that experienced treatment emergent serious adverse events (TESEAs) will be quantified.
Time Frame: 10 - 14 days
Population: Safety Population: all enrolled subjects
Measure: Number; unit: participants
Arm/Group | Treatment Period: 6 mg Triferic IV Over 3 Hours | Treatment Period: 35 Micrograms/kg IV Push
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment Period: 6 mg Triferic IV Over 3 Hours | Treatment Period: 35 Micrograms/kg IV Push
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: 6 mg Triferic IV Over 3 Hours (N=12) | Treatment Period: 35 Micrograms/kg IV Push (N=12)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion Site Swelling (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days